CLINICAL TRIAL: NCT06746285
Title: Artemis: Evaluating the Impact of Synbiotic Supplementation on Infants and Toddlers
Brief Title: Evaluating the Impact of Synbiotic Supplementation on Infants and Toddlers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Persephone Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PB-2024-02
Record Dates: First submitted 2024-12-11; First posted 2024-12-24 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Gastrointestinal Tolerance of Probiotics in Infants
MeSH Terms: interventions — Probiotics; Synbiotics; Lactose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Synbiotic Supplement (Active Comparator): Participants aged 2 months to 24 months will receive daily synbiotic supplementation (probiotic+ prebiotic) for 1 month
  Interventions: Dietary Supplement: Synbiotic Supplement
- Lactose (Placebo Comparator): Participants aged 2 months to 24 months will receive daily placebo (lactose) for 1 month
  Interventions: Dietary Supplement: Lactose (inactive placebo)

INTERVENTIONS:
Dietary Supplement: Synbiotic Supplement — Participants will be given 1g of a synbiotic product each day, containing 4 microbial strains isolated from an infant gut (total of 1 billion cfu) and a mixture of 4 human milk oligosaccharides. Parents will administer the product by dissolving in breast milk, formula, or water, or mixing with food.
  Other Names: probiotic; synbiotic
  Arms: Synbiotic Supplement
Dietary Supplement: Lactose (inactive placebo) — Participants will be given 1g of lactose as a placebo. Parents will administer the product by dissolving in breast milk, formula, or water, or mixing with food.
  Arms: Lactose

SUMMARY:
Background and Significance:

Bifidobacterium longum subspecies infantis (B. infantis) and other infant associated Bifidobacterium (such as Bifidobacterium longum subspecies longum and Bifidobacterium breve) are known to be important bacteria in the infant gut microbiome. A lack of Bifidobacterium in the infant gut may lead to disordered development of the infant microbiome and immune system, which can contribute to the development of gastrointestinal issues, pathogenic infections, and immune-related conditions including allergic disease and autoimmune disorders. The investigators hypothesize that establishing Bifidobacterium in the infant gut through delivery of a synbiotic, containing bifidobacterium and human milk oligosaccharides (HMOs; Bifidobacterium's primary nutrient source) may modulate the microbiome and correct this disruption.

Research Question:

Does synbiotic supplementation on infants and toddlers of various ages alter the gut microbiome as measured by GI-tolerance, fecal microbiome composition, and fecal metabolic profile?

Objectives:

* Demonstrate shifts in microbiome composition and metabolism
* Demonstrate tolerance by observing neutral or positive shifts in GI related behaviors

Study Design Overview:

Participants Infants aged 2-24 months will be enrolled to evaluate the ability of a synbiotic (human milk oligosaccharide + a Bifidobacterium blend (B. infantis, B. longum, and B. breve)) to modulate the gut microbiome. Infants will be randomly split into two cohorts, one that receives synbiotic supplementation and one that receives a placebo control (lactose).

Initially, only ages 12-24 months will be enrolled (first 25 participants), and a safety review will be performed prior to enrolling younger infants.

Cohorts

* Cohort 1 (supplementation) participants will be aged 2 months to 24 months. They will receive synbiotic supplementation for 1 month.
* Cohort 2 (no supplementation) participants will be aged 2 months to 24 months. Will receive placebo (lactose) over the course of 1 month.

Design Caretakers will be recruited and screened using an online questionnaire to determine eligibility and cohort assignment. They will give consent using an online one-party consent form (Appendix 1). Participants will be distributed randomly between cohorts 1 and 2. Participants will be shipped the synbiotic or placebo (lactose) and a set of stool sampling kits. Calls with the participant will take place throughout the study as necessary to explain participant responsibilities and ensure compliance. Two sample types will be collected during the study, a full fecal sample and a DNA/RNA tube only. The full fecal sample will be collected at the beginning and end of supplementation and the DNA/RNA tube only will be collected at all other time points. Samples will be collected at supplementation start, one week after supplementation, four weeks after supplementation start (coinciding with the end of supplementation) and 6 weeks after supplementation start (coinciding with a 2 week washout period). Journals and questionnaires will be used for the duration of supplementation as well as 2 weeks before and after to assess the impact of supplementation.

Laboratory Assessments:

Stool samples will be obtained for each subject. The first sample will be taken before supplementation start. Additional samples will be collected: after 1 week of supplementation, after 1 month of supplementation, and after a 2 week period of no supplementation (a washout period). All samples will be collected at home and shipped back to Persephone Biosciences for processing. The initial sample and the sample after 4 weeks of supplementation will be full samples for metagenomic, metabolomic, and proteomic analysis. The 1 week after supplementation and 2 week post supplementation samples will be DNA/RNA tube samples for metagenomics only. Microbial whole genome sequencing, metabolite analysis, and immune profiling will be performed on stool from complete stool kits. Microbial whole genome sequencing alone will be performed on the DNA/RNA tube kits.

Data Collection:

Demographic data, general health information, diet and lifestyle information will be collected from the subjects (all self-reported). Journals and questionnaires will be used to evaluate the impact of the synbiotic.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of personally signed and dated informed consent document indicating that the caregiver(s) have been informed of all pertinent aspects of the study
2. Caregiver(s) meet the following criteria:

   1. 18 Years or Older
   2. Legal Guardian of the Infant
   3. Intending to cohabitate with the infant/toddler for the duration of the study
   4. Can be reached by phone and email for the duration of the study
   5. Reads, writes, and speaks English
   6. Be able to accurately answer all portions of the questionnaire
   7. Have access to a working freezer
   8. Intending to be primary caregiver and study responder for duration of study
   9. Willing to provide synbiotic either in a bottle or some other format to the infant if on a fully liquid diet
3. The PI considers the Caregiver likely to adequately comply with the study protocol requirements based on demonstrated compliance with initial questionnaires and agreement to complete all diaries
4. The infant or toddler enrolled is:

   1. Healthy (has not been diagnosed with any chronic health conditions by a pediatrician)
   2. Still using diapers (to facilitate sample collection), and expected to continue in diapers for the duration of the study

Exclusion Criteria:

1. Infants/toddlers who have a medical condition or history that could increase the risk associated with study participation or interfere with the interpretation of study results, including:

   * Evidence of major congenital malformations (e.g., cleft palate, extremity malformation)
   * Any history or suspicion of systemic or congenital infections (e.g., human immunodeficiency virus, cytomegalovirus, syphilis)
   * Severe gastroesophageal reflux (throwing up or spitting up more than a teaspoon of milk > 8 times daily)
   * Chronic vomiting (projectile, bilious or bloody emesis)
   * Other severe medical or laboratory abnormality (acute or chronic) which, in the judgment of the investigator, would make the toddler inappropriate for entry into the study
2. Infants/toddlers who are presently receiving or have received within three months prior to enrollment the following:

   * Probiotic supplements
   * Antibiotics
   * Medication(s) or supplement(s) which are known or suspected to affect the following:

     i. fat digestion, absorption, and/or metabolism (e.g., pancreatic enzymes) ii. stool characteristics (e.g., glycerin suppositories, bismuth-containing medications, docusate, Maltsupex, or lactulose) iii. growth (e.g. insulin or growth hormone) iv. gastric acid secretion v. microbiome
3. Infants/toddlers with HIV or hepatitis or lactose sensitivity
4. Infants/toddlers exposed to or displaying symptoms of a disease within 1 month of enrollment, including:

   * Exposure to COVID-19
   * Hematochezia (blood in the stools)
   * Diarrhea (watery stools that takes the shape of a container > 5x daily)
   * Fever (38.2 degrees)
   * Any other symptom which, in the judgment of the investigator, would make the infant inappropriate for entry into the study
5. Currently participating or having participated in another clinical trial since birth

Ages: 2 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate gastrointestinal tolerance of synbiotic supplementation | 1 month
  A modified GIGER index score will be used to determine if there are adverse outcomes related to the synbiotic. This is a scale from 23 to 138, with higher numbers indicating a higher degree of GI discomfort.

SECONDARY OUTCOMES:
Determine impact of supplementation on microbiome composition during intervention | 2 months
  Overall fecal microbiota composition will be assessed using next generation sequencing (NGS) technology. Outcome measure is a list of microbial species and % abundance in each sample, and microbes with differential abundance between the intervention and placebo will be determined.
Determine impact of supplementation on gene function repertoire of the microbiome | 2 months
  Functional genomics will be assessed from the metagenomic sequence data. Metabolic functions with differential abundance between supplementation and placebo will be determined.
Determine rate of probiotic strain colonization | 2 months
  For the participants receiving the synbiotic supplement, a strain-specific microbial classifier will be applied to the sequence data to determine presence of the strains contained in the supplement. For each strain, the fraction of participants in which it is detected will be determined.

CONTACTS AND LOCATIONS:
Locations (1):
- Persephone Biosciences, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be used within the company for trial logistics. Only a limited number of employees, who are involved with stool kit shipping and participant communication, will have access to IPD.

REFERENCES:
- [Background] Pados et al 2021, Global Pediatric Health, 8:1-8